CLINICAL TRIAL: NCT05356715
Title: Bilateral Erector Spinae Plane Block Versus Fentanyl Infusion in Post-operative Recovery in Cardiac Surgery With Median Sternotomy. Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block in Post-operative Recovery in Cardiac Surgery With Median Sternotomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-394-2021
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Sternotomy; Postoperative Pain
Keywords: Erector Spinae; Ultrasound; Sternotomy; Cardiac surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients aged from 18-70 years old, who will undergo open heart surgery procedure through sternotomy will be included in the study. Patients will be randomly allocated into one of two groups:
  * Group A (n=110): will receive Ultrasound guided bilateral ESBP after induction of general anesthesia.
  * Group B (n=110): will receive fentanyl IV infusion 2mic/kg/hr after induction of General anesthesia
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): ● Group A (n=110): will receive Ultrasound guided bilateral ESBP.
  Interventions: Procedure: Ultrasound guided bilateral ESBP
- Group B (Active Comparator): ● Group B (n=110): will receive fentanyl IV infusion 2mic/kg/hr
  Interventions: Procedure: Ultrasound guided bilateral ESBP

INTERVENTIONS:
Procedure: Ultrasound guided bilateral ESBP — Patients in group A will be positioned in the lateral position , ESPB will be done under complete aseptic conditions , using , linear ultrasound probe(Philips HD11XE Ultrasound System) , to locate the ESP at the level of the fifth dorsal vertebrae , 22 G spinal needle will be used to inject 20 ml of 0.25% of bupivacaine in the ESP bilaterally, block will done by an expert anesthesiologist , who will not be included in the data collection

SUMMARY:
This study aim is to measure the time of extubation in patients receiving ultrasound guided bilateral Erector Spinae Plane (ESP) block after cardiac surgery .

DETAILED DESCRIPTION:
On arrival to the operating room, an I.V 20 G cannula will be inserted. . and 500 ml of ringer acetate solution will be infused within 30 minutes. .A five-lead electrocardiogram, a pulse oximeter and an noninvasive blood pressure monitor will be applied. Basal readings ( HR,blood pressur) will be recorded . Then arterial cannula will be inserted in the radial artery of the non dominant hand. Sedation with Midazolam 0.02 mg/kg will be administered at the pre- anethesia room. . Induction will be done using titrated doses of propofol (1-2 mg /kg). ,atracurium 0.5 mg /kg and 200 mcg of fentanyl

* patients will be randomly assigned into two groups :
* Group A (n=110): will receive Ultrasound guided bilateral ESBP.
* Group B (n=110): will receive fentanyl IV infusion 2mic/kg/hr. Patients in group A will be positioned in the lateral position , ESPB will be done under complete aseptic conditions , using , linear ultrasound probe(Philips HD11XE Ultrasound System) , to locate the ESP at the level of the fifth dorsal vertebrae , 22 G spinal needle will be used to inject 20 ml of 0.25% of bupivacaine in the ESP bilaterally, block will done by an expert anesthesiologist , who will not be included in the data collection.

Patients in group B will be on fentanyl infusion 2 mcg /kg/hr. Blood pressure and heart rate will be recorded every 15 min until we go on CPB. An incremental dose of fentanyl bolus 50 mcg will be given when there is increase in the heart rate or the blood pressure by 20% from the baseline. If more than tow boluses needed, then the block will be considered as failed block .Then patients will go on CPB after heparinization and cannulation of the aorta and the venous system ( single venous or double venous ), after valve replacement or CABG done , weaning from the CPB , and inotropic support will start if needed . Then patient will be transferred to ICU mechanically ventilated on assisted control mode, FiO2 :0.6 , TV: 6ml /kg , RR: 12-16/min , PEEP:5. After fulfilling the criteria for extubation ( such as P/F ratio more than 200 , spontaneous tidal volume greater than 5 mL/kg, vital capacity greater than 15 mL/kg, maximum inspiratory pressure (MIP) greater than 25 cm H2O,, fully conscious patient , stable hemodynamics and accepted valves for the arterial blood gases and chest tube drains, patient will be extubated.

All patients will be observed in the postoperative period at 4, 6, 8, 12,24 hours interval and all hemodynamics will be recorded including heart rate ,blood pressure ,the need for incremental doses of narcotics, pain assessment using the Numerical rating scales (NRS), (use numbers to rate pain), and time of extubation ( the time from the arrival to the ICU until successful extubation).

ELIGIBILITY:
Inclusion Criteria:

* patient aged from 18 to 70 years old
* Adult congenital heart disease.
* patients undergoing valve replacement due to valvular heart disease
* Coronary artery bypass grafting( CABG) without great saphenous vein (GSV) harvesting.

Exclusion Criteria:

* Emergency surgeries.
* Allergy to opioids and local anesthetic
* Patients on high inotropic support ( 100 ng/ kg/ min adrenaline or noradrenaline)
* Patients with preoperative known chest disease ( pulmonary function tests showing moderate to severe restrictive or obstructive pulmonary disease
* Long cardiopulmonary bypass (CPB) time ( more than 2 hours )
* Difficult intubation (needs more than 3 attempts bu trained anesthesiologist for a successful endotracheal intubation.)
* Skin lesions or infection at site of proposed needle insertion.
* Bleeding disorders (INR >1.4 ),( platelet count <100,000/mm3 )

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Time to extubation after cardiac surgery | 24 hours
  Time to extubation after cardiac surgery (from the arrival to ICU till successful extubation)

SECONDARY OUTCOMES:
Perioperative fentanyl consumption. | 24 hours
  Perioperative fentanyl consumption.
pain scoring using the Numerical rating scales (NRS) | 24 hours
  pain scoring using the Numerical rating scales (NRS) The NRS consists of a numeric version of the visual analog scale. The most common form of the NRS is a horizontal line with an eleven point numeric range. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Sarhan, MD, Principal Investigator — Lecturer of anesthesia, Cairo university
Locations (2):
- Egypt (2):
  - Cairo university hospitals, kasralainy, Cairo
  - Kasralainy, Cairo

IPD SHARING:
Plan to Share IPD: No